CLINICAL TRIAL: NCT07291232
Title: A Phase 1b Study to Assess the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of Multiple Subcutaneous Doses of ABBV-295 in Adult Subjects With Obesity
Brief Title: A Study of ABBV-295 Subcutaneous Injections to Assess Adverse Events and Pharmacokinetics in Adult Participants With Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M26-089
Record Dates: First submitted 2025-11-19; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Obesity
Keywords: Obesity; ABBV-295
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- ABBV-295 or Placebo-Group 1 (Experimental): Participants will receive subcutaneous doses of ABBV-295 or Placebo for 13 weeks.
  Interventions: Drug: ABBV-295; Drug: Placebo
- ABBV-295 or Placebo-Group 2 (Experimental): Participants will receive subcutaneous doses of ABBV-295 or Placebo for 13 weeks.
  Interventions: Drug: ABBV-295; Drug: Placebo
- ABBV-295 or Placebo-Group 3 (Experimental): Participants will receive subcutaneous doses of ABBV-295 or Placebo for 13 weeks.
  Interventions: Drug: ABBV-295; Drug: Placebo
- ABBV-295 or Placebo-Group 4 (Experimental): Participants will receive subcutaneous doses of ABBV-295 or Placebo for 13 weeks.
  Interventions: Drug: ABBV-295; Drug: Placebo
- ABBV-295 or Placebo-Group 5-Optional (Experimental): Participants will receive subcutaneous doses of ABBV-295 or Placebo for 13 weeks.
  Interventions: Drug: ABBV-295; Drug: Placebo
- ABBV-295 or Placebo-Group 6 (Experimental): Participants will receive subcutaneous doses of ABBV-295 or Placebo for 13 weeks.
  Interventions: Drug: ABBV-295; Drug: Placebo

INTERVENTIONS:
Drug: ABBV-295 — Subcutaneous Injections
Drug: Placebo — Subcutaneous Injections

SUMMARY:
This study is to assess adverse events, change in body weight and pharmacokinetics in adult participants with obesity receiving ABBV-295 subcutaneous injections or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30.0 to ≤ 45.0 kg/m2 after rounding to the tenths decimal at Screening (BMI is calculated as weight in kg divided by the square of height measured in meters) with or without weight related stable comorbidities (e.g., hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease).
* A female who is not pregnant or breastfeeding and is not considering becoming pregnant or donating eggs during the study or for approximately 60 days after the last dose of study treatment.

Exclusion Criteria:

* Participant has a self-reported change in body weight ≥ 5% within 3 months prior to Screening.
* HbA1c ≥ 6.5% and/or serum glucose ≥ 126 mg/dL at Screening.
* Participant has taken a medication for the purpose of treating obesity or has been enrolled in an obesity trial within 180 days prior to study treatment administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 145 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.
Number of Participants with Abnormal Change From Baseline in Vital Sign Measurements | Up to approximately 145 days
  Number of participants with abnormal change from baseline in vital sign measurements like heart rate, systolic and diastolic blood pressure will be assessed.
Number of Participants with Change from Baseline in Electrocardiogram (ECG) | Up to approximately 145 days
  12-lead resting ECG will be recorded.
Number of Participants with Abnormal Change in Clinical Laboratory Test Results Like Hematology will be Assessed | Up to approximately 145 days
  Number of participants with abnormal change in clinical laboratory test results like biochemistry, hematology will be assessed.
Maximum Observed Plasma Concentration (Cmax) of ABBV-295 | Up to approximately 145 days
  Cmax of ABBV-295
Time to Cmax (Tmax) of ABBV-295 | Up to approximately 145 days
  Tmax of ABBV-295
Trough plasma concentration (Ctrough) of ABBV-295 | Up to approximately 145 days
  Ctrough of ABBV-295
Apparent terminal phase elimination rate constant (BETA) of ABBV-295 | Up to approximately 145 days
  BETA of ABBV-295
Terminal phase elimination half-life (t1/2) of ABBV-295 | Up to approximately 145 days
  t1/2 of ABBV-295
Area under the plasma concentration-time curve (AUC) of ABBV-295 | Up to approximately 145 days
  AUC of ABBV-295
Area under the plasma concentration-time curve over the dosing interval (AUCtau) of ABBV-295 | Up to approximately 145 days
  AUCtau of ABBV-295
Dose Normalized Cmax of ABBV-295 | Up to approximately 145 days
  Dose normalized Cmax of ABBV-295 will be assessed.
Dose Normalized AUC of ABBV-295 | Up to approximately 145 days
  Dose normalized AUC of ABBV-295 will be assessed.
Incidence of Anti-Drug Antibodies (ADAs) | Up to approximately 145 days
  Incidence of ADAs will be assessed.
Percent Change in Body Weight From Baseline | Up to approximately 145 days
  Percent change in body weight (kg) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 278624, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M26-089